CLINICAL TRIAL: NCT05869747
Title: Firefighter Collaborative Research Project
Acronym: FCRP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FCRP
Record Dates: First submitted 2023-04-24; First posted 2023-05-22 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-01

CONDITIONS: Exposure; Cardiopulmonary
Keywords: Firefighters
MeSH Terms: interventions — Blood Donation; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Blood Donation (Active Comparator)
  Interventions: Behavioral: Blood Donation; Behavioral: Surveys
- Plasma Donation (Active Comparator)
  Interventions: Behavioral: Plasma Donation; Behavioral: Surveys
- Blood/Plasma Control (Placebo Comparator)
  Interventions: Behavioral: Surveys
- Zone 2 Training (Active Comparator)
  Interventions: Behavioral: Zone 2 Training; Behavioral: Surveys
- Intermittent Fasting (Active Comparator)
  Interventions: Behavioral: Intermittent Fasting; Behavioral: Surveys
- Zone 2 Control (Placebo Comparator)
  Interventions: Behavioral: Surveys
- Intermittent Fasting Control (Placebo Comparator)
  Interventions: Behavioral: Surveys

INTERVENTIONS:
Behavioral: Blood Donation — Participants asked to donate whole blood at a donation facility from a list provided by the study.
  Arms: Blood Donation
Behavioral: Plasma Donation — Participants asked to donate plasma at a donation facility from a list provided by the study.
  Arms: Plasma Donation
Behavioral: Zone 2 Training — Participants asked to work out in their custom Zone 2 heart range 4 times a week for 45 to 60 minutes.
  Arms: Zone 2 Training
Behavioral: Intermittent Fasting — Participants asked to engage in an intermittent fasting routine of a 16 hour fast followed by an 8 hour eating period at least 4 times a week.
  Arms: Intermittent Fasting
Behavioral: Surveys — Participants were asked to complete surveys throughout the study to monitor intervention progress and to collect baseline and end-of-study data.

SUMMARY:
The goal of this research is to test interventions to reduce firefighter cardiovascular, cognitive, and overall disease risks, including but not limited to risks associated with Per- and Polyfluorinated Substances (PFAS) exposure. Approximately 1,500 - 2,000 firefighters will be enrolled in the Fire Fighter Cancer Cohort Study (FFCCS). Among these individuals, those that express interest will then be screened for eligibility for the Firefighter Collaborative Research Project (FCRP) using information they provided for the Fire Fighter Cancer Cohort Study. Firefighters enrolled in the study will provide an initial blood sample and urine sample. The blood sample will be analyzed to determine the participant's PFAS levels. Based upon serum PFAS levels and responses from the screening survey, eligible participants will be randomly assigned into one of the following interventions: 1. Blood Donation, or Plasma Donation or Blood/Plasma Control Group; 2. Zone 2 Training or Zone 2 Control; 3. Intermittent Fasting or Intermittent Fasting Control. Individuals participating in the blood donation, plasma donation or blood/plasma control group would donate blood every 12 weeks, plasma every 6 weeks, or not donate blood or plasma. Participants in this intervention arm would continue this for a 12-month period. Individuals in the zone 2 training, zone 2 training control, intermittent fasting or intermittent fasting control group would participate in their intervention or control for a 4-month period. After 4 to 12 months participating in an intervention or control group, participants will be asked to provide a final urine sample and blood draw to determine if and to what degree their PFAS levels or other cardiovascular disease and other health risks have changed.

ELIGIBILITY:
Inclusion criteria:

* Active firefighter (including emergency medical responder and all firefighter subgroups) with either a volunteer or career status
* Individual plans to remain in active service with their current agency for the next 2 years (not planning to retire or resign)
* 18 years of age and older
* Fluently speak and write in English
* All sexes, races, and ethnicities
* Enrolled in the Fire Fighter Cancer Cohort Study (FFCCS) prior to enrolling in the Firefighter Collaborative Research Project (FCRP)
* Complete a signed and dated informed consent document that indicates the participant has been informed of all aspects of the study prior to enrollment
* Agree to avoid participating in FCRP intervention activities outside of their assigned intervention group for the duration of the study
* Able to comply with scheduled visits, laboratory tests and other study procedures
* BMI of 17.5 kg/m2 or greater and be greater than 115 pounds
* Must also be eligible to donate blood and blood-based products if randomized into the blood or plasmapheresis intervention groups

Exclusion criteria from overall study:

* Not able to fluently speak or write in English
* Less than 18 years of age
* Currently a tobacco smoker or vaping (e.g. >2 cigarettes or cigars, or incidents of vaping in the past month)
* Those with planned travel or extended leave (e.g. >6 weeks) that would prevent their ability to participate in other interventions
* Those who are pregnant, breastfeeding, or have given birth within the past year
* Those with a history or diagnosis of any significant metabolic, hematologic, pulmonary, cardiovascular, gastrointestinal, neurological, immune, hepatic, renal, urological disorders, severe injury or cancer that, in the opinion of the investigator, would potentially put the candidate at risk.

Exclusion criteria from study for those outside of Arizona:

• Those with PFOS levels <5 ng/ml

Exclusion criteria from blood or plasma donation intervention:

* Those with any medical contraindication (medical condition or medication) to blood donation
* Those that donated blood or plasma in the past three months
* Those knowing they have a condition indicative of levels of hemoglobin, hematocrit, red blood cells, or iron below the lower limit of normal levels

Exclusion criteria from the intermittent fasting intervention:

* Those with a history or diagnosis of diabetes, hypoglycemia thyroid disease, and/or an eating disorder
* Those who recently participated in intermittent fasting or Time Restricted Eating
* Those that recently used antidiabetic medication such as Semaglutide (sold as Ozempic, Wegovy, and Rybelsus) or Tirzepatide (sold as Mounjaro) for the treatment of type 2 diabetes or for weight loss will also be excluded from this group.
* Use of drugs that might affect intermittent fasting or eating behaviors
* Those outside of the state of Arizona

Exclusion from the zone-2 physical activity intervention:

* Currently participating in zone 2 physical activity training
* Currently participating in more than 120 minutes per week of aerobic, cardiovascular training (e.g. jogging, cycling, walking, swimming, HIIT) at >60% of their max heart rate.
* Those outside of the state of Arizona or in cities in Arizona where access to CPET testing is not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in concentration of PFAS levels in serum | 12 months
  PFAS levels are per- and polyfluoroalkyl substance levels measured from a biological sample
Change in epigenetic age | 4 months
  Epigenetic age is a mathematically derived age estimators that are based on combinations of methylation values that change with age at specific CpGs in the genome.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Gilbert Fire & Rescue Department, Gilbert, Arizona
  - Green Valley Fire, Green Valley, Arizona
  - Tucson Fire Department Headquarters, Tucson, Arizona
  - Tucson Fire Department Station 9, Tucson, Arizona
  - University of Arizona, Tucson, Arizona
  - Northwest Fire District, Tucson, Arizona
  - Drexel Heights Fire, Tucson, Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Conner R, Porter C, Lutrick K, Beitel SC, Hollister J, Healy O, Kern KJ, Wardenaar F, Gulotta JJ, Jack K, Huentelman M, Burgess JL, Furlong M. Interventions to Reduce Serum Per- and Poly-Fluoroalkyl Substances Levels, Improve Cardiovascular Risk Profiles, and Improve Epigenetic Age Acceleration in US Firefighters: Protocol for Randomized Controlled Trial. JMIR Res Protoc. 2025 Apr 16;14:e67120. doi: 10.2196/67120. PMID 40239196